CLINICAL TRIAL: NCT06285656
Title: Can Femoral Blood Gas Analysis Predict Early Bleeding and the Need for Blood Products After Abdominal Major Surgery: a Prospective Observational Study.
Brief Title: Femoral Blood Gas and Prediction of Postoperative Bleeding
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: ASH-KG
Record Dates: First submitted 2024-02-23; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Hemorrhage; Blood Transfusion
Keywords: Abdominal Surgery; Postoperative Hemorrhage; Blood Transfusion
MeSH Terms: conditions — Postoperative Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Biospecimen Retention: Samples Without DNA — Blood gas
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1/: Patients with postoperative hemmorhagia
- Grup 2: Patients without postoperative hemmorhagia

SUMMARY:
Postoperative bleeding is still an important concern after major abdominal surgery. Postoperative bleeding is the most important determinant of morbidity and death. It results in longer hospital stays, the necessity for extra radiological tests, interventional radiology treatments, and the possibility of reoperation. Early detection of postoperative bleeding reduces morbidity and mortality with appropriate intervention.Simultaneous arterial and venous blood gas measurements can be used to quickly identify the degree of bleeding and the need for replacement in serious trauma patients brought to the emergency room.Lactate levels, venous oxygen saturation, and the differential in partial pressure of carbon dioxide between arterial and venous blood can all be used to indicate the requirement for replacement, as demonstrated in several studies. The purpose of this study is to evaluate lactate levels, venous oxygen saturation, and arterial-venous partial pressure of carbon dioxide difference in blood gas analysis in order to assess the severity of bleeding in patients undergoing major abdominal surgery as early as possible and perform replacement as soon as possible.

ELIGIBILITY:
Inclusion Criteria:

* Patients with major abdominal surgery
* Postoperative intensive care unit following
* Accepting to participate in research

Exclusion Criteria:

* Age under 18 years old
* Pregnant patients
* Do not accept to participate of study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will have surgery at Ankara Bilkent City Hospital's General Surgery Clinic and then be transferred to the critical care unit.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-03 (Estimated)

PRIMARY OUTCOMES:
Eritrocyte replacement | 6 months
  could we predict eritrocyte replacement at early postoperative period?

SECONDARY OUTCOMES:
Postoperative Hemmorhagea | 6 months
  Could we predict postoperative hemorrhage in the early postoperative period?

IPD SHARING:
Plan to Share IPD: No
IPD will not share other researchers.

REFERENCES:
- See also: Femoral blood gas analysis, another tool to assess hemorrhage severity following trauma: an exploratory prospective study — http://sjtrem.biomedcentral.com/articles/10.1186/s13049-023-01095-9
- See also: Prognostic Significance of Blood Lactate and Lactate Clearance in Trauma Patients — https://pubs.asahq.org/anesthesiology/article/117/6/1276/13472
- See also: Changes in central venous saturation after major surgery, and association with outcome — http://ccforum.biomedcentral.com/articles/10.1186/cc3888